CLINICAL TRIAL: NCT05805839
Title: Advanced MR and PET Imaging in Inflammatory Demyelinating Diseases of the Central Nervous System
Brief Title: A Study of Imaging in Demyelinating Diseases
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Burcu Zeydan, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-009149
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Inflammatory Demyelinating Disease
MeSH Terms: conditions — Multiple Sclerosis | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Control Group (Experimental): Subjects without inflammatory-demyelinating diseases of the central nervous system
  Interventions: Drug: C-11 ER176 Radiotracer; Drug: C11 Pittsburgh Compound B; Diagnostic Test: PET/CT scan; Diagnostic Test: MRI
- Multiple Sclerosis Group (Experimental): Subjects with current diagnosis of Multiple Sclerosis or an InflammatoryDemyelinating Disease of the Central Nervous System will have a PET/CT scan with radiotracer drug C-11 PIB & C-11 ER176
  Interventions: Drug: C-11 ER176 Radiotracer; Drug: C11 Pittsburgh Compound B; Diagnostic Test: PET/CT scan; Diagnostic Test: MRI

INTERVENTIONS:
Drug: C-11 ER176 Radiotracer — Administered at a single time IV prior to the PET imaging. The injected dose of C-11 ER176 will be 518 MBq (14 mCi) (range 370-666 MBq; 10-18 mCi).
Drug: C11 Pittsburgh Compound B — Administered at a single time IV prior to the PET imaging. The injected dose of C-11 PiB will be 555 MBq (range 370 - 629 MBq).
Diagnostic Test: PET/CT scan — Imaging of entire brain
Diagnostic Test: MRI — Magnetic Resonance Imaging of the Brain

SUMMARY:
This purpose of this study is research the usefulness of MRI with PET/CT imaging for measuring brain inflammation and its relation to Multiple Sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Meet the requirements for one of the case or control groups.
* MS patients undergoing neurologic evaluation procedures as part of Understanding Sex Differences in Multiple Sclerosis Spectrum of Demyelinating Disorders (IRB# 19-002807) Study or the Mayo Clinic Neurology Multiple Sclerosis Clinic.
* Control participants without inflammatory-demyelinating diseases of the central nervous system
* Capacity to sign consent.

Exclusion Criteria:

* Participants unable to lie down without moving for 20 minutes.
* Women who are pregnant or cannot stop breast feeding for 24 hours.
* For all patients and controls, any acute glucocorticoid (e.g., IV methylprednisolone or PO prednisolone) use within 2 weeks is an exclusion to limit medication interaction but preserve possible chronic systemic inflammation interaction with microglia activation metrics. Chronic disease modifying treatments in MS are allowed as these medications are not known to impact microglia activation.
* Standard safety exclusionary criteria for MRI such as metallic foreign bodies, pacemaker, etc., since the quantitative PET data analysis is based on anatomic criteria that are established uniquely for each subject by registration to his/her MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Uptake of C-11 Pittsburgh compound-B (PiB) in white matter myelin | Baseline
  C-11 Pittsburgh compound-B (PiB) in PET imaging measured by PiB standardized uptake value ratio (SUVr)
Uptake of C-11 ER176 Radiotracer | Baseline
  C-11 ER176 Radiotracer in TSPO PET imaging measured by ER176 SUVr

SECONDARY OUTCOMES:
Number of subjects with adverse events | 2 days
  Total number of subjects to experience adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Zeydan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials